CLINICAL TRIAL: NCT05934422
Title: Nutritional Intervention Preconception and During Pregnancy to Maintain Healthy Glucose Metabolism and Offspring Health - Child Health and Well-being Follow Up Study
Brief Title: NiPPeR Randomised Trial - Child Follow Up Study
Acronym: NiPPeR Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National University Hospital, Singapore (Other); Auckland UniServices Ltd. (Industry); Institute for Human Development and Potential (IHDP), Singapore (Other); National University of Singapore (Other); National University Health System, Singapore (Other); University of Auckland, New Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 79093
Record Dates: First submitted 2023-05-04; First posted 2023-07-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Childhood; Cognition; Neurobehavioral Manifestations; Metabolic Disturbance; Growth Disorders; Allergy; Atopic Dermatitis; Atopy; Nutrition, Healthy; Lifestyle; Microbial Colonization; Breastfeeding
Keywords: Nutrition; Body composition; Neurodevelopment; Lifestyle; Endocrinology and metabolism; Preconception; Supplementation; Pregnancy; Infancy; Breast milk
MeSH Terms: conditions — Pediatric Obesity; Neurobehavioral Manifestations; Growth Disorders; Hypersensitivity; Dermatitis, Atopic; Communicable Diseases; Breast Feeding | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prior Intervention - enhanced micronutrients, probiotics, myo-inositol in preconception & pregnancy (Experimental): NiPPeR Study intervention drink containing a mix of micronutrients, probiotics and myo-inositol given to the mother during preconception & pregnancy
  Interventions: Other: Intervention (Study Nutritional Drink)
- Prior Control - standard micronutrients in preconception & pregnancy (Active Comparator): NiPPeR Study control nutritional drink containing a mix of micronutrients given to the mother during preconception & pregnancy
  Interventions: Other: Control (Standard Nutritional Drink)

INTERVENTIONS:
Other: Intervention (Study Nutritional Drink) — Study nutritional drink containing a mix of enriched micronutrients, probiotics and myo-inositol.
  Arms: Prior Intervention - enhanced micronutrients, probiotics, myo-inositol in preconception & pregnancy
Other: Control (Standard Nutritional Drink) — Control nutritional drink containing a standard mix of micronutrients
  Arms: Prior Control - standard micronutrients in preconception & pregnancy

SUMMARY:
There is an increasing focus on the need to optimise nutrition, lifestyle and metabolism of parents before and during pregnancy and of the infant after birth, but as yet there is limited understanding of the specific influences and of the underlying mechanisms.

This study is a follow up of children from the NiPPeR trial of a nutritional drink enriched with micronutrients, myo-inositol and probiotics taken preconception and during pregnancy. In this setting we will examine the influence of parental nutrition, lifestyle and metabolism before and during pregnancy on child growth, development and well-being; ascertaining growth, adiposity, metabolism, neurobehavioural and health outcomes in the children, and characterising the underlying mechanisms.

The data collected will allow identification of the contributions of parental and offspring characteristics, nutritional, lifestyle and medical factors, social and economic status, ethnicity, genetics, metabolism and microbes to promoting healthy growth, body composition and wellbeing in the children.

ELIGIBILITY:
Inclusion Criteria:

All children still participating in the NiPPeR study at 6-8 years.

Exclusion Criteria:

Known significant congenital anomaly or genetic condition that influences child growth or neurodevelopment.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 461 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Child Body Mass Index (kg/m2), derived from weight and height | Up to age 8 years, from periconception to age 8 years
  Child size and body composition
Intellectual function (WASI-II IQ [4 sub-test scores], higher score is a higher IQ) | Up to age 8 years, from periconception to age 8 years
  Child cognition
Child insulin resistance (HOMA2-IR [no units], higher value is greater insulin resistance) | Up to age 8 years, from periconception to age 8 years
  Child insulin resistance
Dimensional Change Card Sort Test (raw & T-scores) | Up to age 8 years, from periconception to age 8 years
  Child executive functioning - NIH Toolbox Cognition Battery component
Flanker Inhibitory Control & Attention Test (raw & T-scores) | Up to age 8 years, from periconception to age 8 years
  Child executive functioning - NIH Toolbox Cognition Battery Component
Strengths & Difficulties Questionnaire score (no units) | Up to age 8 years, from periconception to age 8 years
  Child neurobehavioural functioning
Child Behaviour Check List score (no units) | Up to age 8 years, from periconception to age 8 years
  Child neurobehavioural functioning

SECONDARY OUTCOMES:
Body fat mass (kg, % and indices) | Up to age 8 years, from periconception to age 8 years
  Obesity and body composition
Change in body fat mass (kg) | Up to age 8 years, from periconception to age 8 years
  Adiposity gain
Body lean mass (kg, % and indices) | Up to age 8 years, from periconception to age 8 years
  Child body composition - lean mass
Change in lean mass (kg) | Up to age 8 years, from periconception to age 8 years
  Lean mass gain
Body bone mass (kg, % and indices) | Up to age 8 years, from periconception to age 8 years
  Child body composition - bone mass
Change in bone mass (kg) | Up to age 8 years, from periconception to age 8 years
  Bone mass gain
Child height (cm) | Up to age 8 years, from periconception to age 8 years
  Child height
Height growth (cm) | Up to age 8 years, from periconception to age 8 years
  Linear growth
Change in body mass index (z-score & percentile) | Up to age 8 years, from periconception to age 8 years
  Change in BMI
Change in weight (kg) | Up to age 8 years, from periconception to age 8 years
  Weight gain
Child mid-upper arm circumference (cm) | Up to age 8 years, from periconception to age 8 years
  Child arm circumference
Change in mid-upper circumference (z-score) | Up to age 8 years, from periconception to age 8 years
  Change in soft tissue mass
Child waist circumference (cm) | Up to age 8 years, from periconception to age 8 years
  Child waist circumference
Change in waist circumference (z-score) | Up to age 8 years, from periconception to age 8 years
  Adiposity gain
Heart rate response to step test (beats per minute) | Up to age 8 years, from periconception to age 8 years
  Cardiovascular fitness and function
Child blood pressure (mm Hg) | Up to age 8 years, from periconception to age 8 years
  Cardiovascular fitness and function
Child resting heart rate (beats per minute) | Up to age 8 years, from periconception to age 8 years
  Cardiovascular fitness and function
Child minutes to return to resting heart rate (minutes) | Up to age 8 years, from periconception to age 8 years
  Cardiovascular fitness and function
Diagnosed medical conditions or disorders ascertained by questionnaire, including child medical conditions, infections, gastrointestinal, cardiovascular, respiratory, dermatological, neuropsychological, mental and musculoskeletal health and wellbeing | Up to age 8 years, from periconception to age 8 years
  Child health and wellbeing
Dietary patterns ascertained by frequency questionnaires | Up to age 8 years, from periconception to age 8 years
  Child diet
Child Eating Behaviour Questionnaire | Up to age 8 years, from periconception to age 8 years
  Child eating behaviours
Parental Feeding Practices Questionnaire | Up to age 8 years, from periconception to age 8 years
  Parental feeding practices
Children's Sleep Habits Questionnaire | Up to age 8 years, from periconception to age 8 years
  Child sleep patterns
Children's actigraphy measurements of activity behaviours [minutes/day] | Up to age 8 years, from periconception to age 8 years
  Child physical activity, sleep and sedentary behaviours
Child Movement Behaviour Questionnaire | Up to age 8 years, from periconception to age 8 years
  Child activity behaviours
Skin pricks test results to allergens [mm] | Up to age 8 years, from periconception to age 8 years
  Child atopic sensitisation
Child asthma, wheezing illnesses, eczema, rhinitis and food allergy by clinical examination & questionnaires | Up to age 8 years, from periconception to age 8 years
  Child atopic and allergic wellbeing and disorders
Hair metabolome panel concentrations (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Biomarkers of health and wellbeing measured in hair samples
Urine micronutrient concentrations (nmol/L) | Up to age 8 years, from periconception to age 8 years
  Child micronutrient status
Blood micronutrient concentrations (nmol/L) | Up to age 8 years, from periconception to age 8 years
  Child circulating micronutrient profile
Blood trace element concentrations (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child circulating trace element profile
Urine trace element concentrations (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child trace element status
Stool metagenomic profile (abundance) | Up to age 8 years, from periconception to age 8 years
  Child gut microbiota composition
Skin metagenomic profile (abundance) | Up to age 8 years, from periconception to age 8 years
  Child skin microbiota composition
Stool metatranscriptomic profile (relative activity) | Up to age 8 years, from periconception to age 8 years
  Child gut microbiota activity profile
Skin metatranscriptomic profile (relative activity) | Up to age 8 years, from periconception to age 8 years
  Child skin microbiota activity profile
Stool metabolomic profile (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child gut microbiota metabolite profile
Skin metabolomic profile (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child skin microbiota metabolite profile
Blood molecular profile (% methylation) | Up to age 8 years, from periconception to age 8 years
  Child blood epigenetic profile
Buccal molecular profile (% methylation) | Up to age 8 years, from periconception to age 8 years
  Child buccal cell epigenetic profile
Blood transcriptomic profile (relative expression) | Up to age 8 years, from periconception to age 8 years
  Child blood transcriptomic profile
Buccal transcriptomic profile (relative expression) | Up to age 8 years, from periconception to age 8 years
  Child buccal cell transcriptomic profile
Genetic variation (DNA sequence analysis) | Up to age 8 years, from periconception to age 8 years
  Genetic variant analysis
Circulating chemocytokine measurements (nmol/L) | Up to age 8 years, from periconception to age 8 years
  Child chemocytokine profile
Circulating adipokine measurements (nmol/L) | Up to age 8 years, from periconception to age 8 years
  Child adipokine profile
Circulating inflammatory marker measurement (nmol/L) | Up to age 8 years, from periconception to age 8 years
  Child inflammatory factor profile
Plasma glucose concentration (mmol/L) | Up to age 8 years, from periconception to age 8 years
  Child's plasma glycemia
Plasma lipid concentrations (mmol/L) | Up to age 8 years, from periconception to age 8 years
  Child's metabolic profile - lipid concentrations
Plasma high-sensitivity C-reactive protein concentrations (mmol/L) | Up to age 8 years, from periconception to age 8 years
  Child's inflammatory marker status
Blood metabolome panel concentrations (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child's blood metabolomic status
Urine metabolome panel concentrations (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Child's urine metabolomic status
Urine measurement of environmental pollutant exposure (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Urine exposome pollutant profile
Blood measurement of environmental pollutant exposure (ng/gm lipid) | Up to age 8 years, from periconception to age 8 years
  Blood exposome pollutant profile
Hair measurement of environmental pollutant exposure (pmol/L) | Up to age 8 years, from periconception to age 8 years
  Hair exposome pollutant profile

OTHER OUTCOMES:
Healthcare utilisation (US$) | Up to age 8 years, from periconception to age 8 years
  Health economics analysis of child outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Wayne S Cutfield, MB MD FRACP, Principal Investigator — The University of Auckland; Shiao-Yng Chan, MD PhD FRCOG, Principal Investigator — National University of Singapore; Keith M Godfrey, BM PhD FRCP, Principal Investigator — MRC Lifecourse Epidemiology Centre, University of Southampton
Locations (3):
- The University of Auckland, Auckland, New Zealand
- National University Hospital, Singapore, Singapore
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godfrey KM, Cutfield W, Chan SY, Baker PN, Chong YS; NiPPeR Study Group. Nutritional Intervention Preconception and During Pregnancy to Maintain Healthy Glucose Metabolism and Offspring Health ("NiPPeR"): study protocol for a randomised controlled trial. Trials. 2017 Mar 20;18(1):131. doi: 10.1186/s13063-017-1875-x. PMID 28320484
- [Background] Godfrey KM, Barton SJ, El-Heis S, Kenealy T, Nield H, Baker PN, Chong YS, Cutfield W, Chan SY; NiPPeR Study Group. Myo-Inositol, Probiotics, and Micronutrient Supplementation From Preconception for Glycemia in Pregnancy: NiPPeR International Multicenter Double-Blind Randomized Controlled Trial. Diabetes Care. 2021 May;44(5):1091-1099. doi: 10.2337/dc20-2515. Epub 2021 Mar 29. PMID 33782086